CLINICAL TRIAL: NCT05172115
Title: Catheter-Directed Thrombolysis Versus ANticoagulation Monotherapy in Patients With Acute Intermediate-High Risk PulmonarY Embolism: The CANARY Randomized Clinical Trial
Brief Title: Catheter-Directed Thrombolysis Versus Anticoagulation Monotherapy in Intermediate-High Risk PE
Acronym: CANARY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Responsible Party: Principal Investigator, Parham Sadeghipour, Associate Professor, Rajaie Cardiovascular Medical and Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 97056
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Pulmonary Embolism; Pulmonary Thromboembolisms; Embolism, Pulmonary; Right Ventricular Dysfunction
Keywords: Intermediate-high risk pulmonary embolism; Catheter-directed thrombolysis; Anticoagulation
MeSH Terms: conditions — Pulmonary Embolism; Ventricular Dysfunction, Right | interventions — carbohydrate-deficient transferrin; Enoxaparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: 1:1 open-label parallel group randomized controlled trial with concealed allocation sequence and blinded outcome adjudication
Who Masked: Outcomes Assessor
Masking Description: Allocation sequence concealment and blinded outcome adjudication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional catheter-directed thrombolysis (CDT) (Experimental): Conventional catheter-directed thrombolysis (CDT) will be the interventional arm. CDT will be administered using fixed-dose of 24 mg tissue plasminogen activator infusion over 24 hours (0.5 mg/h per catheter if bilateral or 1 mg/h per unilateral catheter) with 500 unit per hour of infusion of unfractionated heparin during the thrombolytic therapy. The therapeutic dose of heparin will immediately be substituted the CDT after termination, and twice-daily subcutaneous enoxaparin (1mg/kg) for the first 48 hours after the thrombolytic therapy will be administered. Direct oral anticoagulation will be in ones with no clinical deterioration.
  Interventions: Procedure: Conventional catheter-directed thrombolysis (CDT) with recombinant tissue plasminogen activator (rtPA)
- Anticoagulation-only therapy (Active Comparator): The anticoagulation-only therapy will be the assigned treatment in the control arm. Control patients will receive subcutaneous enoxaparin (twice-daily, 1mg/kg) in the first 48hours of enrollment. Direct oral anticoagulation will be in ones with no clinical deterioration.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Procedure: Conventional catheter-directed thrombolysis (CDT) with recombinant tissue plasminogen activator (rtPA) — Conventional catheter-directed thrombolysis with fixed-dose of 24 mg tissue plasminogen activator infusion over 24 hours
  Other Names: Cragg-McNamara™ valved infusion catheters
  Arms: Conventional catheter-directed thrombolysis (CDT)
Drug: Enoxaparin — Subcutaneous enoxaparin twice-daily (1mg/kg)
  Other Names: low molecular weight heparin (LMWH)
  Arms: Anticoagulation-only therapy

SUMMARY:
In an open-label parallel groups blinded-endpoint randomized clinical trial, the investigators aim to assess the safety and efficacy of conventional catheter-directed thrombolysis (CDT) vs anticoagulation monotherapy on outcomes of patients with acute intermediate-high risk pulmonary embolism. The investigators hypothesize that CDT will have a superior efficacy and safety compared with anticoagulation-only therapy regarding the proportion of patients with a right ventricle to left ventricle (RV/LV) ratio > 0.9 at a 3-month follow-up by an imaging core laboratory, major bleeding, severe thrombocytopenia, or vascular access complication.

DETAILED DESCRIPTION:
Treatment of intermediate risk PE is still debated. Despite the promising results of small studies on the efficacy and safety of systemic thrombolytic therapy, larger trials failed to show a net clinical benefit. Pulmonary EmbolIsmTHrOmbolysis (PEITHO) trial which compared the full-dose systemic thrombolysis (i.e., tenecteplase) versus anticoagulation therapy in patients with intermediate-risk PE showed significant lower incidence of mortality or hemodynamic collapse in the first 7 days after randomization in patients who received tenecteplase (2.6% vs 5.6% in placebo group, [odds ratio, 0.44; 95% confidence interval, 0.23 to 0.87; P value, 0.02]). However the mortality benefit was neutralized by the increased risk of major bleeding in thrombolytic arm (11.5% vs 2.4% in the tenecteplase and placebo group, respectively. Importantly, during the long-term follow up (median of 37.8 months) of PEITHO participants, the thrombolytic therapy failed to improve the RV right ventricular function, residual dyspnea ( 36% in thrombolysis group vs 30.1% in the placebo group), or mortality rates (20.3% in thrombolysis group vs 18 % in the placebo group ). CTEPH occurred in ( 2.1% in thrombolysis group vs 3.2% in the placebo group. The lack of benefit of full-dose thrombolytic in PEITHO, might have several explanations. Intermediate risk PE compose of heterogenous group of patients with different prognosis in whom one fits all approach would not be applicable. This heterogeneity in prognosis were underlined in the latest guideline of the European Society of Cardiology (ESC) which classified the intermediate-risk PE category into two groups of intermediate-low and intermediate-high risk patients according to the right ventricle function and cardiac biomarker levels. Second, lower-dose thrombolytic regimen might result in the same benefit with lower bleeding events. CDT, by delivering drug locally, claims to increase the efficacy of thrombolytic agents and consequently decrease the required dose which might translate to lower bleeding events.

In an open-label parallel groups blinded-endpoint randomized clinical trial, we aim to evaluate the safety and efficacy of standard catheter-directed thrombolysis (CDT) vs anticoagulation-only therapy in patients with acute intermediate-high risk pulmonary embolism. The hypothesis is that CDT will have a superior efficacy and safety regarding the proportion of patients with a RV/LV ratio > 0.9 at a 3-month follow-up assessed by an imaging core laboratory with the lower complications of major bleeding, severe thrombocytopenia, and vascular access complication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years
2. Confirmed acute pulmonary emboli by computed tomography pulmonary angiography (CTPA)
3. Symptom onset ≤14 day
4. Elevated N-terminal-proB-type natriuretic peptide and cardiac troponin
5. Right ventricle/left ventricle ratio >0.9 in transthoracic echocardiography
6. Less than 48 hours of anticoagulation therapy
7. Willingness for participation in the study with signed and dated informed consent form

Exclusion Criteria:

1. Pulmonary emboli detected by modalities other than CTPA
2. Segmental PE
3. High risk (massive)
4. Severe renal dysfunction(creatinine clearance [CrCl] below 30 mL/min)
5. Terminal illness Surgery within 2 weeks
6. Platelet count <50.000 /µL
7. Pre and post catheter directed thrombolysis echocardiography exam not possible
8. Contraindication to thrombolytic therapy
9. Concomitant right heart thrombi
10. Allergic reaction to study medications
11. Lack or withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-12-22 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a RV/LV ratio >0.9 | At 3 months from randomization
  Proportion of patients with a RV/LV ratio >0.9 at a assessed by an imaging core laboratory 3-month follow-up

SECONDARY OUTCOMES:
The proportion of patients with an RV/LV ratio >0.9 | At 72 hours from randomization
  A composite of the proportion of patients with a RV/LV ratio >0.9 at a assessed by an imaging core laboratory 72 hours follow-up
The proportion of patients with Unrecovered RV | At 3 months from randomization
  The PEITHO definition for RV recovery was employed, as follows: 1) RV size (at the mid-cavity level In apical 4-chamber view) <35 mm, 2) pulmonary artery pressure <35 mm Hg, 3) an RV/LV ratio <0.9, and 4) the normalization of RV free wall motion. The fulfillment of all the criteria, some criteria, and none of the criteria was defined as complete, partial, and no recovery, respectively.
All-cause mortality | Within 3-month Study period
  Survival status of the patient (being alive or dead) at the end of 3 months follow up
Major bleeding | Within 3-month Study period
  According to the Bleeding Academic Research Consortium (BARC 3 or 5 bleeding)
Severe thrombocytopenia | Within 3-month Study period
  Platelet count <20.000/µL
Vascular access complication | Within 3-month Study period
  Major vascular access complication

OTHER OUTCOMES:
A composite of all-cause death or the primary outcome | Within 3-month Study period
  Composite patients who died or patients with a RV/LV ratio >0.9 at a assessed by an imaging core laboratory 3-month follow-up
PE-related mortality. | Within 3-month Study period
  Autopsy-confirmed PE with no more likely cause of death or objectively confirmed PE before death in the absence of another more likely cause of death
Hospital length of stay | Within 3-month Study period
  The total days of the initial hospitalization
Six-minute walk test (6MWt) at three-month follow up | Within 3-month Study period
  The functional capacity of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Parham Sadeghipour, M.D, Principal Investigator — Rajaie Cardiovascular Medical and Research Center
Locations (1):
- Rajaie Cardiovascular Medical and Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
Data will become available to interested investigators upon submitting a reasonable research request, approved by the Steering Committee of the trial.

REFERENCES:
- [Derived] Sadeghipour P, Jenab Y, Moosavi J, Hosseini K, Mohebbi B, Hosseinsabet A, Chatterjee S, Pouraliakbar H, Shirani S, Shishehbor MH, Alizadehasl A, Farrashi M, Rezvani MA, Rafiee F, Jalali A, Rashedi S, Shafe O, Giri J, Monreal M, Jimenez D, Lang I, Maleki M, Goldhaber SZ, Krumholz HM, Piazza G, Bikdeli B. Catheter-Directed Thrombolysis vs Anticoagulation in Patients With Acute Intermediate-High-risk Pulmonary Embolism: The CANARY Randomized Clinical Trial. JAMA Cardiol. 2022 Dec 1;7(12):1189-1197. doi: 10.1001/jamacardio.2022.3591. PMID 36260302